CLINICAL TRIAL: NCT04538417
Title: Cooled Radiofrequency Ablation for the Treatment of Refractory Phantom and Residual Limb Pain; a Pilot Study.
Brief Title: C-RFA of Residual Limb Neuroma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Zachary McCormick, MD FAAPMR, Associate Professor, Director of Clinical Spine Research, Director of Interventional Spine and Musculoskeletal Medicine Fellowship, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 106250
Record Dates: First submitted 2020-08-28; First posted 2020-09-04 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Phantom Limb Pain; Neuroma Amputation
Keywords: Cooled Radiofrequency Ablation
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: Participants who meet inclusion and exclusion criteria will be enrolled into the study after consenting to participate and before receiving residual limb neuroma C-RFA. This procedure is considered standard of care and are typically based on physician preference. Data will be collected by questionnaire at baseline and select follow up timelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Residual Limb Pain in affected amputated limb (Other): Patient has residual limb pain in amputated limb and is scheduled to receive standard of care treatment of cooled radiofrequency ablation.
  Interventions: Device: Cooled Radiofrequency Ablation

INTERVENTIONS:
Device: Cooled Radiofrequency Ablation — RFA procedures will be performed with modification accounting for appropriate C-RFA technique. Participant will be positioned prone and skin prepped with chloroprep. Ultrasound probe will be placed on residual limb at a transverse angle in order to view the nerve and associated neuroma in long-axis. The probe will be advanced to the site of the stump neuroma. C-RFA electrode will be placed adjacent to neuroma. Needle will be connected via wire to a cooled radiofrequency generator. Motor and sensory testing will be performed to reproduce or exacerbate the RLP and / or PLP. At the site of the neuroma, 2 mL of local anesthetic will be injected through the needle. C-RFA lesions will be created by using the typical C-RFA protocol. Upon completion needle will be removed. Following ablation, 0.5 mL of 0.5% bupivacaine will be injected at the site of the ablated neuroma to provide post procedure analgesia.

SUMMARY:
To assess changes in pain, physical function, and health-related quality of life in patients with post-amputation neuroma-associated residual limb pain after cooled radiofrequency ablation.

DETAILED DESCRIPTION:
Residual limb (RLP) and phantom limb pain (PLP) affects most amputees at some point in their life1. The incidence of PLP has been estimated to range between 50 - 80%. RLP prevalence has been estimated to be 43%. The peak of onset is bimodal and often appears within the first month and second year after amputation. RLP is more common in the first year after amputation, with PLP becoming the predominate amputee pain complaint after one-year post-amputation.

Both RLP and PLP fall under the umbrella term "post-amputation pain." While these conditions are frequently found in combination, their clinical features and underlying causes are distinct. PLP is a painful sensation in the distribution of the missing limb. Following amputation, abnormalities at multiple levels of the neural axis have been implicated in the development of PLP; changes include cortical reorganization, reduced inhibitory processes at the spinal cord, synaptic response changes and hyperexcitability at the dorsal root ganglion, and retrograde peripheral nerves shrinkage.

Residual limb pain has been called "neuroma pain" and is mechanistically distinct from PLP11. Neuromas may form as early 6-10 weeks after nerve transection, and are thought the produce ectopic neural discharges resulting in severe pain. Evidence suggests RLP and PLP commonly co-occur and patients may struggle to differentiate between these pain types. Risk factors include female sex, upper extremity amputation, pre-amputation pain, residual pain in contralateral limb, and time since amputation.

Depression, anxiety, and stress are known to exacerbate PLP / RLP. Patients experiencing PLP and RLP also experience a higher incidence of indecisiveness, suicidal ideation, and thoughts of self-harm8. Current guidelines for treatment of PLP and RLP are not standardized. Treatments includes pre-operative analgesia, neuromodulation mirror therapy, imagery, acupuncture, transcranial stimulation, deep brain stimulation, and medications (including, but not limited to: TCAs, SSRIs, gabapentinoids, sodium channel blockers, ketamine, opioids, and NSAIDs). Many agents have been injected in neuromas. These include local anesthetic, phenol, alcohol, and botulinum toxin. These oral, intravenous, and nonpharmacological modalities have demonstrated limited success in the treatment of PLP / RLP. Neuroma cryoablation has been used, but this method of neural destruction poses technical challenges related to cumbersome needle placement and the requirement for time-intensive freeze-thaw cycles.

Conventional RFA has been studied on RLP. Zhang et. al treated 13 patients with painful stump neuromas. The study started with alcohol neurolysis before using ultrasound-guided RFA for refractory cases. The frequency of sharp pain was reduced in all RFA-treated patients. Kim et. al described a case in which ultrasound-guided RFA was successfully used to treat a sciatic neuroma of an above-knee amputee.

No outcome literature on the effectiveness of C-RFA technology has been published. C-RFA is similar in mechanism to conventional RFA: a thermal lesion is created by applying radiofrequency energy through an electrode placed at a target structure. In C-RFA, a constant flow of ambient water is circulated through the electrode via a peristaltic pump, maintaining a lowered tissue temperature by creating a heat sink. By removing heat from tissues immediately adjacent to the electrode tip, a lower lesioning temperature is maintained, resulting in less tissue charring adjacent to the electrode, less tissue impedance and more efficient heating of target tissue. The volume of tissue heated, and the resultant thermal lesion size is substantially larger with C-RFA, conferring an advantage over conventional RFA. Further, given the spherical geometry and forward projection the C-RFA lesions beyond the distal end of the electrode, the RFA probe can be positioned at a range of possible angles and still capture the target neural structure, whereas more fastidious, parallel positioning is required with conventional RFA. These technical advantages increase the probability of successful denervation of neural pain generators that have variability in anatomic location. Additionally, a longer lesion of the RLP-generating nerve may be more reliably achieved with C-RFA compared to conventional RFA.

As such, the present study aims to define the attributable effect of cooled RFA on pain, physical function, and health-related quality of life in patients with post-amputation neuroma-associated residual limb pain. This prospective single-arm pilot study is intended to inform a future properly powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years of age at day of enrollment.
2. Clinical diagnosis lower extremity amputation performed more than 1 year since study enrollment.
3. Residual pain described as burning pain and sensations of movement in the affected amputated limb32.
4. Pain duration of more than 6 months despite a trial of conservative therapy (medications, physical therapy) for 2 months.
5. Ultrasound and / or MRI imaging pathology consistent with clinical symptoms and signs.
6. Greater than 50% pain relief with a diagnostic neuroma block

Exclusion Criteria:

1. Refusal or inability to participate, provide consent, or provide follow-up information for the 12-month duration of the study.
2. Contraindications to diagnostic block or treatment ablation (active infection, bleeding disorders, and pregnancy or breastfeeding, active immunosuppression, participation in another phantom or residual limb pain trial within the last 30 days
3. Non-neurogenic source of residual or phantom limb pain.
4. Active moderate to severe lumbar radiculopathy.
5. Any injection in the residual limb within the last 30 days.
6. Severe uncontrolled medical condition as determined by treating physician.
7. Severe psychological illness.
8. History of Inflammatory arthritis.
9. Malignancy within past 5 years except basal cell or squamous cell skin cancer. 10. Current opioid use exceeding50morphinemilligram equivalents per day.

11. A history of alcohol or drug abuse within past 5 years. 12. Use of any investigational drug within past 30 days. 13. Pending litigation involving participant's residual limb pain. 14. Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Residual Limb Pain in Affected Amputated Limb
Started | 8
Withdrew to Have Phenol Ablation | 1
Withdrew to Have Targeted Muscle Reinnervation Therapy | 1
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Residual Limb Pain in Affected Amputated Limb
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 60.3 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7
Height [Mean (Standard Deviation); unit: Centimeters] | 166.2 (16.17)
Weight [Mean (Standard Deviation); unit: Kilograms] | 86.8 (19.17)
Duration of Pain [Count of Participants; unit: Participants]
  < 1 Year | 1
  1 to 5 Years | 4
  > 5 Years | 2

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) for Pain at 6 Months
Description: Presented here is the proportion of participants reporting ≥50% improvement in Numeric Rating Scale pain score at 6 months after their cooled radiofrequency ablation procedure. The Numeric Rating Scale was used to quantify neuroma-associated residual limb pain by asking patients to rate their pain intensity on an 11-point scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Residual Limb Pain in Affected Amputated Limb
Number analyzed (Participants) | 7
Participants | 4

2. Secondary Outcome: Median Change in Numeric Rating Scale (NRS) Scores for Pain
Description: Patients rated their residual limb pain intensity at baseline and the designated follow-up timepoints using an 11-point Numeric Rating Scale (NRS) ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable". Change scores were calculated by subtracting follow-up scores from baseline scores. Median change scores and their interquartile ranges are reported here. Positive median change scores indicate pain improvement from baseline, with greater values corresponding to greater pain relief. Similarly, negative change scores indicate worsening pain from baseline.
Time Frame: 1, 3, 6, and 12 months
Population: Of the 7 participants included in the analyses, one participant withdrew from the study after outcome data were collected at 6-month follow-up to pursue alternative treatment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Residual Limb Pain in Affected Amputated Limb
Number analyzed (Participants) | 7
units on a scale
  1 month | 1.0 [0.5 to 3.0]
  3 months | 2.0 [1.5 to 2.5]
  6 months | 1.0 [-1.5 to 3.0]
  12 months: number analyzed (Participants) | 6
  12 months | 3.0 [1.3 to 4.0]

3. Secondary Outcome: Medication Quantification Scale III Mean Score
Description: The Medication Quantification Scale (MQS) is calculated using a pain-related medication detriment score based on drug class, which ranges from 1.1 to 4.5, and multiplying it by a usage score: 1 = subtherapeutic or occasional dose/2 = lower 50% of a therapeutic dose/ 3 = upper 50% of a therapeutic dose/ 4 = supratherapeutic dose. The higher the score, the more pain-related medication the participant takes to control their pain. The resulting score is useful in research for tracking individual or group pain medication use over time.
Time Frame: 1, 3, 6 and 12 Months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Residual Limb Pain in Affected Amputated Limb
Number analyzed (Participants) | 7
Score on a scale
  1 Month | 8.3 [6.1 to 10.0]
  3 Months | 6.9 [4.6 to 8.1]
  6 Months | 7.1 [3.6 to 8.5]
  12 Months: number analyzed (Participants) | 6
  12 Months | 7.1 [2.4 to 9.7]

4. Secondary Outcome: Proportion of Patients With a ≥6 Score on Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change is a scale which measures participant reported satisfaction after an intervention. The outcome was measured as the percent of patients reporting a PGIC score of 6-7 (indicating "much improved" and "very much improved").
Time Frame: 1, 3, 6, and 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Residual Limb Pain in Affected Amputated Limb
Number analyzed (Participants) | 7
Participants
  1 month | 3
  3 months | 3
  6 months | 1
  12 months: number analyzed (Participants) | 6
  12 months | 1

ADVERSE EVENTS:
Time Frame: The day of the procedure
Description: The only adverse events that will be documented are those that occurred immediately after ablation and are related to the procedure.
Arm/Group | Residual Limb Pain in Affected Amputated Limb
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04538417/Prot_SAP_000.pdf